CLINICAL TRIAL: NCT05177250
Title: The Possible Association Between Bisphenol A, Paraben Exposure and Type 2 Diabetic Adult Patients.
Brief Title: Association of Bisphenol A,Paraben Exposure and Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Fathy Hussein Awad, Assistant lecturer of forensic medicine and clinical toxicology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: bisphenol A,paraben, type 2DM
Record Dates: First submitted 2021-12-09; First posted 2022-01-04 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Type2 Diabetes; Bisphenol A
MeSH Terms: interventions — Chromatography, High Pressure Liquid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Other): 50 cases with type 2 DM.
  Interventions: Device: HPLC
- Control group (Other): 50 subjects not diabetics.
  Interventions: Device: HPLC

INTERVENTIONS:
Device: HPLC — taking urine samples from participants and analyze these samples to detect bisphenol A and paraben

SUMMARY:
The aim of this study is to evaluate the association between BPA , paraben levels and type 2 DM patients

DETAILED DESCRIPTION:
The first phase of the study will include a questionnaire :

* The cases and control will be asked about demographic information such as residence, age, education, and occupation.
* History of discovery of diabetes.
* Exposure to products and materials such as polycarbonate plastics, cosmetics and beverages containing bisphenol A and paraben and it will be evaluated through exposure sheet through asking about dietary exposure, Environmental exposure and medical exposure.

Then clinical evaluation including:

* Full clinical examination will be performed for cases and control.
* Anthropological data:

their weights, heights and waist circumference will be measured. The body mass index (BMI) will be calculated by weight (kg)/height (m)2 formula.

* Investigations: routine and specific investigation as blood glucose level, HbA1c and lipid profile.
* Urine specimens will be collected in clean, glass containers will labeled with the subject identification number. Turbid sample or those containing blood will be excluded.
* All specimens will be stored frozen below 20 degree centigrade.
* Urine samples will be analyzed by High Performance liquid chromatograph (HPLC) to detect bispenol A and parabens levels.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ( 18 y or elder).
2. Type 2 DM

Exclusion Criteria:

* Type 1 DM
* Less than 18 y
* History of chronic diseases such as liver failure, cardiac patients……etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Bisphenol A and paraben detection in urine samples of diabetic (n=50) and non diabetic persons (n=50) | Baseline
  Evaluation of bisphenol A and Paraben detection in urine samples from type 2 diabetic adult patients compared with non diabetic persons using HPLC

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Fathy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No